CLINICAL TRIAL: NCT04960852
Title: Color Match Assessment of a Single Shade Structurally Colored Universal Resin Composite: A Single Arm Clinical Trial
Brief Title: Color Match Assessment of a Single Shade Structurally Colored Universal Resin Composite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Shaymaa Mohamed Nagi, Assisstant professor in restorative and dental materials department, National Research Centre, Egypt
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3433042021
Record Dates: First submitted 2021-07-02; First posted 2021-07-14 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Dental Caries (Disorder)
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- a single shade structurally colored universal resin composite (Experimental): Cavities will be prepared. one shade universal composite (Omnichroma) a will be applied according to the manufacturer.
  Interventions: Other: a single shade structurally colored universal resin composite

INTERVENTIONS:
Other: a single shade structurally colored universal resin composite — Omnichroma is a single shade composite that is claimed to have blending effect with the tooth color, thus eliminate shade matching procedures during restorative treatment

SUMMARY:
Matching the color of resin composite utilized in anterior teeth is believed to be one of the most challenging tasks a dentist has to face in daily practice. The color of the teeth is primary influenced by dentin; on the other hand, enamel has a major influence on the color perception in terms of lightness. In the layering concept, the missing dental tissues are substituted in increments with resin composite of the exact shade as the dental tissue. A translucent composite resin is applied over a more opaque composite resin to achieve a depth perception similar to that of the natural teeth. Which indicates that the visible color is the consequence of diffuse reflectance from the internal dentin or opaque material layer through the external translucent layer.

There are numerous elements that make the color matching problematic. These problems arise from the point that color matching rely on many different chromatic properties related to the teeth and resin composite; those include hue, chroma and value; translucency, opalescence and fluorescence; light diffusion and transmission; and luster and texture of the surface. To reach the ideal esthetics, restorative material should mimic the natural tooth in the previously mentioned properties, in addition of having a long time color stability.

Massive efforts were achieved over the years to improve the esthetic properties of dental resin composite restorative materials. Recently, a single shade structurally colored universal composite (Omnichroma, Tokuyama Dental) intended for use with most direct restorative clinical cases was introduced in the market. Its manufacturer claimed that it exhibits color change toward the color of the surrounding hard dental tissues. Thus, it has the advantages of improving the esthetic appearance of the restoration, decrease dependence on shade-matching procedures, decrease the number of shade guide tabs, and counteract for color mismatches to some degree.

Up till now no studies assessed the color match of Omnichroma resin composite in anterior teeth cavities clinically. Thus, the aim of this clinical trial was to investigate if the single shade structurally colored universal resin composite (OMNICHROMA) will modify its shade to match the tooth structure shade in anterior teeth cavities.

DETAILED DESCRIPTION:
Participants' recruitment:

The patients will be selected from outpatient clinic of National Research Centre (NRC), Cairo; Egypt Eligible patients who agreed to participate in this trial will sign on written informed consents.

Clinical procedure

* Teeth color measurement Each patient first will receive scaling and polishing procedures to clean the teeth surfaces. A total of 45 anterior teeth cavities will be prepared. Before cavity preparation, shade determination will be performed with Vita Easyshade spectrophotometer. The probe tip will be positioned perpendicular and flushed onto the buccal surface of the tooth to get correct measurements.
* Cavities preparation Appropriate local dental anesthesia (Mepecaine-L) 1mg will be injected preoperatively unless declined by the patient. Treated teeth will be properly isolated and saliva ejector will be utilized.

Conservative cavities will be prepared with #330 carbide bur (FG, Dentsply Midwest®) fixed to a high speed hand piece with water coolant system. Cavity preparation will be limited to the removal of caries and the exact cavity form and size will be obtained after caries removal. Each bur will be discarded after 5 preparations.

A functional esthetic enamel bevel will be prepared using a fine grained finishing diamond rotary instrument on the facial surface, the bevel enables harmonious shade transition from composite to tooth substance.

- Application of the adhesive system and resin composite in the prepared cavities Enamel of the prepared cavities will be etched using UltraEtch (Ultradent, 40% phosphoric acid) for 30 seconds. After rinsing with water and air drying, the bonding agent will be applied according to the manufacturer's instructions to the cavity using a brush then air-thinned gently and light-cured for 20 seconds.

Omnichroma resin composite will be packed in the prepared cavities using a Teflon coated plastic instrument and the restoration will covered with celluloid strip to reduce the oxygen inhibition layer and to get a smooth surface, then light-cured for 40 sec. Excess material will be removed with scalpel. Finishing and polishing will be performed for the anatomical contouring and smoothing of the restorations surfaces using all grates of soflex discs, fine and Extra fine diamond burs, medium and fine rubber polishing points.

Color assessment Color match data will be recorded for the restoration after one week. The restorations will be gently dried with cotton and the color values of them will be recorded using the Vita Easyshade spectrophotometer.

The color changes (ΔE) will be calculated from the changes in CIE L, a, and b values (ΔL, Δa, Δb) as follows:

ΔE= [(ΔL)2 + (Δa)2 + (Δb)2]1/2 CIE Lab is expressed by the L coordinate representing color luminosity, varying from white to black, a and b coordinates representing the chromaticity of the color, with axes varying from green to red and blue to yellow, respectively. The mean of the values obtained will be calculated, and the L, a, and b parameters will be determined.

Visual assessment Visual assessment will be performed by two independent observers with normal color vision as checked by Ishiara test. To determine the color-matching between the restorations and the teeth. Color-matching visual scoring (VS) values will be expressed numerically as follows: 1: mismatch/totally unacceptable, 2: Poor-Match/hardly acceptable, 3: Good- Match/acceptable, 4: Close-Match/small-difference, and 5: Exact-Match/no-color-difference. All observers will be trained in color-matching and taught about the used grading system before the assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with carious class V or Class III cavities
* Young adult Males or female
* patient with low or moderate caries risk index
* Co-operative patients approving to participate in the study

Exclusion Criteria:

* Patients with a compromised medical history
* Severe or active periodontal disease
* Severe medical complications
* Erosive lesions
* Lack of compliance and rampant caries

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-08-06 (Actual); Study Completion 2021-08-06 (Actual)

PRIMARY OUTCOMES:
shade matching (digital analysis) | after 1 week of restorations placement
  to assess the shade matching of the newly introduced OMNICHROMA resin composite to the tooth structure. Image analysis will be carried out by comparing LAB values using Easyshade spectrophotometer

SECONDARY OUTCOMES:
shade match acceptance (visual assessment) | after 1 week of restorations placement
  shade match acceptance will be evaluated by two observers Color-matching visual scoring (VS) values will be expressed numerically as follows: 1: mismatch/totally unacceptable, 2: Poor-Match/hardly acceptable, 3: Good- Match/acceptable, 4: Close-Match/small-difference, and 5: Exact-Match/no-color-difference.

CONTACTS AND LOCATIONS:
Overall Officials: Shaymaa M Nagi, pHD, Principal Investigator — National Research Centre, Egypt
Locations (1):
- National research centre, Cairo, Egypt

REFERENCES:
- [Background] Ragain JC, Johnston WM. Color acceptance of direct dental restorative materials by human observers. Color Res Appl. 2000;25(4):278-285. Riad MI, Gamal WM, Morsy AS. Color matching of a single shade structurally colored universal resin composite with the surrounding hard dental tissues. Egyptian Dental Journal; 2020, 66, 2721:2727. Kim BJ, Lee YK. Influence of the shade designation on the color difference between the same shade-designated resin composites by the brand. Dent Mater. 2009;25: 1148-54. Mohamed MA, Afutu R, Tran D, Dunn K, Ghanem J, Perry R and Kugel G. Shade-Matching Capacity of Omnichroma in Anterior Restorations. J Dental Sci 2020, 5(2): 000247. Kevin B. How to match any composite restoration shade: Tokuyama's OMNICHROMA Uses Smart Chromatic Technology to Match a Wider Range of Natural Teeth Colors. Dental Products Report 2019; 53(3): 36.